CLINICAL TRIAL: NCT05528653
Title: Telehealth as a Modality to Increase the Uptake of PrEP Services in Black and Latino: "e-PrEP"
Acronym: e-PrEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vivent Health (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Cindy Firnhaber, Principal Investigator, Vivent Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IN-US-412-6419
Record Dates: First submitted 2022-05-19; First posted 2022-09-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: HIV Prevention
Keywords: HIV
MeSH Terms: interventions — emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Descovy (Other): Descovy for PrEP
  Interventions: Drug: Descovy

INTERVENTIONS:
Drug: Descovy — HIV infection pre-exposure prophylaxis

SUMMARY:
To evaluate if utilizing Telehealth medicine for access to HIV PrEP will engage more Black and Latino Men who have sex with Men (MSM)

DETAILED DESCRIPTION:
The goal of this study is to determine whether incorporating a telehealth model that allows for same-day appointments for PrEP delivery with the support of navigation leads to increased uptake and persistence of PrEP in young MSM/transgender of color and individuals in rural communities that have disproportionately not used PrEP. The investigators will accomplish this by using an effectiveness-hybrid design that will allow us to both evaluate the interventions impact on relevant clinical outcomes as well as the effectiveness of the implementation strategy. Our hypothesis is that by removing some of the barriers to care such as transportation, childcare, work schedule and potentially stigma with repeated clinic visits, the investigators will increase the uptake and persistence of PrEP amongst communities who historically have had many barriers to care and have not started PrEP.

ELIGIBILITY:
Inclusion Criteria:

1. HIV negative on any FDA approved HIV test within 10 days of starting PrEP 18 years and older
2. No medical or mental health comorbidity that would preclude participating in a clinical study as deemed by the study investigator
3. Able to understand and sign consent in English or with other language interpreter
4. Able to stay in the state catchment area of the license health care provider
5. No use of PrEP for more than 30 days in the last year

Exclusion Criteria:

1. HIV positive
2. If greater and equal to 50 years of age and Renal Glomerular Filtration Rate (GFR) <30 mg/g
3. <18 years of age
4. No access to Internet or devise for telehealth
5. Cis-gender Women

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
: To increase the number and proportion of individuals who start PrEP who have been under-represented in PrEP uptake including those who identify as Black and/or Latino MSM. | 18 months
  Offer PrEP care via tele-health to reduce obstacles that clients have in coming to clinic.

SECONDARY OUTCOMES:
To increase the number and proportion of individuals who are still taking PrEP and engaged in care at the end of 6 months by 30% and remain HIV negative including those who identify as Black and/or Latino MSM. | 18 months
  Facilitate maintenance of care by offering Tele-health for initial and ongoing PrEP care to reduce social and structural barriers.
To assess the acceptability and implementation of the intervention by both patients and clinic staff. | 18 months
  Obtain quantitative feedback via survey about services provided via Telehealth from patients and clinic staff.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Firnhaber, MD, Principal Investigator — Vivent Health
Locations (3):
- United States (3):
  - Vivent Health, Denver, Colorado
  - Vivent Health, St Louis, Missouri
  - Viventh Health, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No